CLINICAL TRIAL: NCT01058616
Title: Phase 1 Dose-escalation Study of LTX-315 in Patients With a Transdermally Accessible Tumour
Brief Title: Dose-escalation Study of LTX-315 in Patients With a Transdermally Accessible Tumour
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Collaborators: Oslo University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C08-315-01
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Cancer With Transdermal Accessible Tumour
MeSH Terms: interventions — LTX-315

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: LTX-315 (Oncopore™) — 5 mg/ml-70 mg/ml. Dosing will be done as transdermal injection of a calculated volume at day 1 and 8. Additionally weekly injections up to a maximum of 4 injections.

SUMMARY:
The study will evaluate the safety profile for LTX-315 a lytic-peptide that has shown effect in animal models to kill cancer tumours when injected directly in to the tumour. The study will also monitor the immunological response in the body after injection of LTX-315.

DETAILED DESCRIPTION:
A phase I study with an initial concentration/volume escalating part followed by an expanded cohort at the recommended dose (RD). This is an open label, multicentre study assessing the safety, tolerance, PK and efficacy of LTX-315 injected directly into transdermally accessible tumours on days 1 and 8.

Additional weekly injections may be made, for up to a total of 6 injections.

Subjects may be included in the study if they meet all of the following criteria:

1. Histologically confirmed malignant tumour
2. Transdermally accessible lesion (in or close to the skin)
3. Age ≥ 18 years
4. ECOG Performance status (PS): 0 - 2
5. Life expectancy: At least 3 months

The primary objectives of the study are to evaluate the safety profile of LTX-315 by assessment of adverse events and abnormal laboratory values recorded during the study and to determine the recommended dose of LTX-315.

The secondary objectives of the study are to preliminarily assess the anti-tumour activity of LTX-315 in patients with transdermally accessible tumours, monitor immunological response, pharmacokinetic assessment, and determine duration of response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant tumour. Transdermally accessible lesion (in or close to the skin) of 1 - 5 cm in diameter.
* ECOG Performance status (PS): 0 - 2
* Life expectancy: At least 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Evaluate safety profile of LTX-315 by assessment of adverse events and abnormal laboratory values recorded during the study. Necrosis of the target tumour based on imaging and core biopsy analysis. | 12 weeks

SECONDARY OUTCOMES:
Assessment of the anti-tumour activity: Objective response in the target tumour, response in non-target tumours, Immunological response. | 12 weeks
Core biopsy staining for lymphocyte infiltratio | 12 weeks
Tumour volume measurment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paal Brunsvig, MD, PhD, Principal Investigator — Oslo University Hospital, Radiumhosptalet, Oslo, Norway
Locations (2):
- Oslo University Hospital, Radiumhospitalet, Oslo, Norway
- Karolinska University Hospital, Solna, Stockholm, Sweden